CLINICAL TRIAL: NCT05188170
Title: Phase 1 Study of Niclosamide (ANA001) in Pediatric Patients With Relapsed and Refractory AML
Brief Title: Niclosamide in Pediatric Patients With Relapsed and Refractory AML
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: The Leukemia and Lymphoma Society (Other); Pediatric Cancer Research Foundation (PCRF) (Unknown); CURE Childhood Cancer, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-61916; PEDSHEMAML0007 (Other: OnCore); 641095 (Other Grant/Funding Number: CURE Childhood Cancer); 6587-20 (Other Grant/Funding Number: Leukemia & Lymphoma Society); NCI-2022-09974 (Registry Identifier: National Cancer Institute Clinical Trials Reporting Program)
Record Dates: First submitted 2021-11-30; First posted 2022-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Niclosamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Niclosamide 250 mg/m2 /day divided BID (Experimental)
  Interventions: Drug: Niclosamide
- Niclosamide 500 mg/m2 /day divided BID (Experimental)
  Interventions: Drug: Niclosamide
- Niclosamide 800 mg/m2 /day divided BID (Experimental)
  Interventions: Drug: Niclosamide
- Niclosamide 1200 mg/m2 /day divided BID (Experimental)
  Interventions: Drug: Niclosamide

INTERVENTIONS:
Drug: Niclosamide — Niclosamide will be administered orally for 14 days. Each dose will be followed by backbone chemotherapy

SUMMARY:
Protocol is designed to evaluate a niclosamide dose escalation scale in combination with cytarabine as a therapeutic modality for pediatric subjects with relapsed/refractory acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. Prior morphologically-confirmed diagnosis of AML based on WHO Criteria 2. Has previously failed all available and suitable therapies for AML. Disease relapse or the presence of refractory disease after ≥ 2 cycles of intensive chemotherapy; or ≥ 4 cycles of non-intensive chemotherapy or hypomethylating agents (HMAs) must be documented by bone marrow (BM) examination demonstrating ≥ 5% blasts in the BM by morphology or ≥ 1% blasts by flow cytometry,

* 5% blasts in the peripheral blood (confirmed by flow cytometry, cytogenetics or FISH), ≥ 1% MRD

  + by flow cytometry, FISH, PCR or NGS, and not attributable to another cause (EXCEPTION: subjects with frank disease progression in the face of treatment with HMA with or without venetoclax will be considered eligible regardless of treatment cycles administered if they meet the other eligibility criteria). No prior treatment with niclosamide. 3. Age ≥ 2 and ≤ 30 years 4. Body surface area (BSA) ≤ 2.10 m2

  , calculated per the Mostellar formula 5. Must be able to tolerate po or ng medications. 6. Performance status: Subject ≤ 16 years old: Lansky ≥ 50 Subject > 16 years old: Karnofsky ≥ 50% 7. Life expectancy of greater than 4 weeks 8. Platelets ≥ 10,000/mm3 (for subjects with platelets < 10,000/mm3 at baseline, platelet transfusion support is allowed) 9. Measured or calculated creatinine clearance
* 60 mL/min/1.73 m2 (by the Cockcroft-Gault method) within 14 days prior to treatment initiation 10. Total bilirubin ≤ 2.0 x institutional upper limit of normal (ULN) within 14 days prior to treatment initiation (EXCEPTION: Subjects with Gilbert's syndrome may be included if the total bilirubin is

  * 3.0 x ULN) 11. SGOT (AST) ≤ 3.0 x ULN and SGPT (ALT)
  * 3.0 x ULN within 14 days prior to treatment initiation 12. Patients must have received their last dose of anti-cancer therapy (chemotherapy, immunotherapy, targeted agents, radiotherapy or investigational therapy) at least 2 weeks or 3 half-lives prior to the start of study treatment, whichever is longer. 13. For patients who have received prior hematopoietic stem cell transplants (HSCT), no evidence of GvHD and must be > 60 days since the HSCT. HSCT recipients must have completed their last course of tacrolimus, cyclosporine, or mycophenolate > 4 weeks before initiation of niclosamide 14. Females of reproductive potential (WOCBP) must have a negative pregnancy test within 14 days prior to study treatment. WOCBP must agree to use adequate contraception (eg, hormonal or barrier methods of birth control; abstinence; sterilized partner) from date of consent through the treatment period, and for 30 days after completion of niclosamide administration 15. Men only: Men must agree to use adequate contraception (eg, hormonal or barrier methods of birth control; abstinence; sterilized partner) from date of consent through the treatment period, and for 30 days after completion of niclosamide administration 16. Ability to understand the purpose and risks of the study and the willingness to sign a written informed consent document containing an authorization to use protected health information (in accordance with national and local subject privacy regulations

Exclusion Criteria:

1. Received anticancer therapy (chemotherapy, immunotherapy, radiotherapy, or investigational therapy) within 2 weeks prior to starting study treatment. Administration of hydroxyurea 10 to 20 mg/kg/day PO (maximum 1000 mg PO BID) to control high WBC > 50 x 103

   /mm3 is permitted at MD discretion (however, hydroxyurea should be stopped at least 24 hours prior to protocol therapy start).
2. Receiving any other investigational agents, including niclosamide.
3. Unresolved toxicities due to prior anticancer therapy, defined as not having resolved to Grade 0 or 1 (by CTCAE version 5 criteria), unless otherwise defined in the inclusion/exclusion criteria with the exception of alopecia
4. Acute promyelocytic leukemia (French-American-British Class M3-AML)
5. Known active central nervous system (CNS) leukemia; subjects can enroll on study if CNS disease can be cleared with intrathecal chemotherapy, in the judgement of the treating physician
6. Known congenital bleeding disorders, including but not limited to hemophilia
7. Known active uncontrolled systemic infection
8. Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, uncontrolled symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction, at the time of study entry
9. Inability to receive administration of niclosamide in the available formulation(s)
10. Uncontrolled intercurrent illness including, but not limited to, uncontrolled active infection, or psychiatric illness/social situations that would limit compliance with study requirements
11. Lactating or pregnant female
12. Known active hepatitis C

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | 30 days
  Dose-limiting toxicities (DLTs) are defined as any events ≥ Grade 3 that are at least possibly, probably, or definitely related to niclosamide treatment

SECONDARY OUTCOMES:
Efficacy of niclosamide treatment clinical response | 8 weeks
  Clinical response is defined as any of the following.
  * Complete response (CR) = < 5% blasts in BM, with no evidence of extramedullary disease.
  * Partial response (PR) = ≥ 5% to ≤ 25% blasts in BM with decrease in BM blast percentage by 50%, and no evidence of extramedullary disease.
  * Resistant disease with clinical benefit (RD-CB) = either ≥ 5% to ≤ 25% blasts in BM OR a decrease in blast percentage by 50%, either with no evidence of extramedullary disease.
  No response (NR) is defined as BM disease that does not fall into the above categories

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Sakamoto, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No